CLINICAL TRIAL: NCT05749055
Title: The ENCALM Trial: A Randomized, Double-blind, Placebo-controlled Monotherapy Trial to Evaluate the Efficacy and Safety of ENX-102 in Patients With Generalized Anxiety Disorder
Brief Title: ENCALM: A Study of ENX-102 as a Monotherapy Treatment in Patients With Generalized Anxiety Disorder
Acronym: ENCALM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Engrail Therapeutics INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENX-102-003
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ENX-102 (Experimental): Four weeks of 2 mg of ENX-102 in capsule form followed by 3 weeks of tapered dose plus 2 weeks of placebo in capsule form (before and/or after the ENX-102 treatment period), taken orally once daily in the evening for a 9-week total treatment period.
  Interventions: Drug: ENX-102
- Placebo (Placebo Comparator): Nine weeks of placebo in capsule form taken orally once daily in the evening for a 9-week total treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ENX-102 — Selective GABA-A alpha2,3,5 positive allosteric modulator
  Arms: ENX-102
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The ENCALM trial is designed to evaluate the efficacy and safety of ENX-102 in patients diagnosed with generalized anxiety disorder (GAD)

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female at birth, inclusive of any gender identity, aged 18 to 65 years, inclusive, at Screening
* Diagnosed with GAD according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), confirmed by a Mini-International Neuropsychiatric Interview (MINI) version 7.0.2
* Experiencing clinically significant generalized anxiety in need of treatment as measured by Hamilton Anxiety Rating Scale (HAM-A) Screening and Day 1 scores ≥22 and at least moderately severe score symptoms of anxious mood and tension as measured by HAM-A items 1 and 2, respectively, with score each ≥2 at Screening and Day 1

Key Exclusion Criteria:

* Clinically predominant psychiatric diagnosis other than GAD as confirmed by the MINI
* Any past/lifetime/current diagnosis of a neurocognitive disorder, or psychotic disorder, or any current diagnosis of posttraumatic stress disorder, obsessive compulsive disorder or bipolar disorder confirmed by independent adjudication
* Reports moderately severe to severe symptoms of depression
* Ingested psychotropic medication within 5 half-lives or 21 days (whichever is longer) prior to Day 1, including THC and CBD, and unwillingness to refrain from their use for the entire duration of the trial
* Recent suicidal ideation or behavior
* Current or recent moderate to severe substance use disorder as assessed by the MINI
* Clinically significant abnormal findings in safety assessments
* Has significant progressive disorders or unstable medical conditions
* Unable to comply with the requirements of the study or, in the opinion of the Investigator or Sponsor, is unsuitable for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of ENX-102 versus placebo in patients with generalized anxiety disorder (GAD) | 4 weeks
  Mean change from baseline on the Hamilton Anxiety Rating Scale (HAM-A) total score [14 symptoms with each symptom scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56 and higher scores representing worse outcomes]

CONTACTS AND LOCATIONS:
Overall Officials: Estibaliz Arce, PhD, Study Director — Engrail Therapeutics INC
Locations (32):
- United States (32):
  - IMA Clinical Research Phoenix, Phoenix, Arizona
  - Collaborative Neuroscience Research, LLC (CNS), Garden Grove, California
  - Sun Valley Research Center, Imperial, California
  - Alliance Research, Long Beach, California
  - NRC Research Institute, Los Angeles, California
  - Excell Research, Inc., Oceanside, California
  - Anderson Clinical Research, Redlands, California
  - California Neuroscience Research, LLC, Sherman Oaks, California
  - Pacific Clinical Research Management Group, Upland, California
  - Sunwise Clinical Research, Walnut Creek, California
  - Mountain View Clinical Research, Denver, Colorado
  - Vertex Clinical Research, Clermont, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Accel Research Sites Network - Lakeland CRU, Lakeland, Florida
  - Accel Research Sites Network - Maitland CRU, Maitland, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - CenExel iResearch, LLC, Savannah, Georgia
  - Collective Medical Research, Overland Park, Kansas
  - Boston Clinical Trials, Boston, Massachusetts
  - Precise Research Centres, Flowood, Mississippi
  - IMA Clinical Research, Las Vegas, Nevada
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Neurobehavioral Research, Cedarhurst, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Austin Clinical Trials Partners, Austin, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Aim Trials, Plano, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Alpine Research Organization, Clinton, Utah
  - Core Clinical Research, Everett, Washington

IPD SHARING:
Plan to Share IPD: No